CLINICAL TRIAL: NCT04887662
Title: The Effects of Regular Consumption of Fermented Vegetables on the Gut Bacteria and Markers Associated With Cardiovascular Disease in Overweight Adults
Brief Title: Happy Gut Study - Fermented Vegetables and Cardiovascular Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1712254-1
Record Dates: First submitted 2021-05-04; First posted 2021-05-14 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Cardiovascular Diseases
Keywords: C-reactive protein; lipopolysaccharide binding protein; trimethylamine oxide; Oxidized LDL receptor
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will be asked to follow their usual diet, but will receive print materials about a diet for cardiovascular health.
- Fermented vegetable (Experimental): The fermented vegetable group will be asked to consume 100 g of fermented vegetables per day, at least 5 days per week for 8 weeks.
  Interventions: Other: Fermented vegetable

INTERVENTIONS:
Other: Fermented vegetable — Participants will be asked to consume 100 g of fermented vegetables per day, at least 5 days per week, for 8 weeks
  Arms: Fermented vegetable

SUMMARY:
The purpose of this project is to determine whether regular consumption of fermented vegetables can decrease inflammation and change the types of bacteria that are normally present in the large intestine. Recent research studies have linked the gut bacteria to many disorders and conditions, such as obesity, cardiovascular disease, diabetes, etc. We also know that certain bacteria are considered probiotic bacteria because they contribute to a healthy gut, while others have been associated with inflammation and disease. Fermented foods may contain beneficial bacteria that may improve health in humans. However, there is a lack of research studies examining the effects of regular consumption of fermented foods on health. This study will help investigators better understand if regular consumption of fermented vegetables can improve inflammation and change the gut bacteria towards a more beneficial profile.

DETAILED DESCRIPTION:
Investigators will recruit 90-100 participants for this study. Participants will be recruited by posting flyers throughout Jacksonville, social media advertisements, and by advertisements on public radio. Recruitment flyers and advertisements will direct potential participants to email or call study staff or visit the study website. The study website will direct potential participants to answer the screening questions and those found to be eligible will be asked to provide contact information so that study staff can contact them to schedule an orientation via zoom. The study orientation will last approximately 45 minutes and will include a PowerPoint presentation about the study, outlining all procedures and a thorough review of the consent form.

After the study orientation, participants will be given two weeks to contact the study if they wish to participate. Those who decide to participate will be asked to schedule their baseline appointment by calling or emailing the study. During the initial appointment, participants will be asked to sign a copy of the consent form and any additional questions they might have about the study will be answered. Both the baseline and follow up visits will take place in building 39/39A, 3rd floor. The time frame between the orientation and the baseline appointment will range between 2 and 3 weeks.

Procedures prior to each clinic visit

There will be a total of two clinic visits, and the same procedures apply to both:

Once participants schedule their first visit, they will be mailed a stool collection kit containing three collection tubes, a collection hat, and a liner for the collection hat, along with instructions on how to collect the stool samples. These instructions will also be available on the study's website. These samples will be collected prior to the first clinic visit, so that participants can bring the collection tubes with them to the clinic visit.

Participants will also be sent information on how to fill out online questionnaires and they will be asked to complete the questionnaires prior to their clinic visit. The questionnaires will ask about demographic information, medical history, diet history and physical activity. The study website will contain all the data collection materials, so that enrolled participants can easily access these documents. Every randomized participant will receive a password to the website to access the study's materials.

Procedures during each clinic visit The two clinic visits will take approximately 45 minutes, each and they will be scheduled in the morning hours, because participants will have to fast for 12-hours to provide blood samples. Participants will be greeted by study staff and their temperature will be checked as part of the covid screening. Then, they will be taken to the body composition assessment lab, for measurement of weight, height, and body fat % using the InBody 570. Participants will be asked to stand on a platform and hold on to the handles of the equipment for approximately 2 minutes for the assessment of body composition. Next, participants' blood pressure will be measured twice using a digital blood pressure monitor and they will be asked to recall their food consumption over the past 24 hours(24-hr diet recall). Lastly, trained nurses will collect approximately 16 mL of blood in two tubes.

At the first clinic visit, participants randomized into the treatment group will receive print materials about a heart-healthy diet and a four-week supply of fermented vegetables with a measuring cup for easy portioning of the vegetables. They will also be asked to fill out an electronic symptoms log where they will list any side effects associated with food consumption, weekly. Participants randomized to the control group will only receive print materials about a heart-healthy diet, but they will also be asked to fill out the symptoms log.

Following the first clinic visit, participants will be contacted by study staff once a week by phone or text-message, depending on their preferred method of contact. The weekly checks will serve to remind participants to fill out the symptoms log and to check on compliance in the case of the treatment group, by asking participants if they skipped any days or consumed less vegetables than prescribed for the week. At four weeks, all participants will be asked to provide another 24-hr diet recall, and another four-week supply of fermented vegetables will be delivered to participants in the treatment group.

Data collection All questionnaire data will be filled out electronically with the exception of the three 24-hr recalls that will be done in person or by phone. All questionnaire data will be identified with a unique ID number that will be assigned to each participant. There will be only one file that will include participants' name with ID numbers, which will be password protected and stored in a secured drive.

ELIGIBILITY:
Inclusion Criteria:

* BMI over 25.9
* Generally healthy

Exclusion Criteria:

* Diabetes
* Taking statins
* Taking monoamine oxidase inhibitors
* Salt sensitivity
* Uncontrolled hypertension
* Diagnosed with Autoimmune disease
* Regular use of probiotics
* Regular use of antibiotics
* Pregnant or breastfeeding

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Change in C-reactive protein | baseline and 8 weeks later
  ng/mL
Change in oxidized LDL receptor | baseline and 8 weeks later
  pg/mL
Change in trimethylamine oxide | baseline and 8 weeks later
  ng/mL
Change in lipopolysaccharide binding protein | baseline and 8 weeks later
  ng/mL
Change in Shannon Index | baseline and 8 weeks later
  no unit

SECONDARY OUTCOMES:
Change in angiopoietin-like protein 4 | baseline and 8 weeks later
  ng/mL

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website — http://www.happygut.domains.unf.edu

DOCUMENTS (1):
  • Informed Consent Form (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT04887662/ICF_000.pdf